CLINICAL TRIAL: NCT02933320
Title: A Cancer Research UK Phase I/IIa Clinical Trial of BI-1206; an Antibody to FcƔRIIB (CD32b), as a Single Agent and in Combination With an Anti-CD20 Antibody in Patients With CD32b Positive B-cell Malignancy
Brief Title: BI-1206 and an Anti-CD20 Antibody in Patients With CD32b Positive B-cell Lymphoma or Leukaemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Collaborators: BioInvent International AB (Industry); Bloodwise (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRUKD16001; 2015-004999-29 (EudraCT Number)
Record Dates: First submitted 2016-09-26; First posted 2016-10-14 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: B-cell Lymphoma; Chronic Lymphocytic Leukaemia; Waldenström Macroglobulinemia
Keywords: Indolent B-cell Lymphoma; Chronic Lymphocytic Leukaemia; Waldenström Macroglobulinemia; BI-1206; CD32b
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, B-Cell; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: Arm 1: BI-1206 single agent dose escalation phase (Experimental): BI-1206 given by IV infusion to all patients once weekly for a period of four weeks, patients will then have a follow-up period of four weeks (8 week period classified as induction therapy).
  Interventions: Biological: BI-1206 single agent dose escalation phase
- Part A: Arm 2: Combination of BI-1206 with rituximab escalation phase (Experimental): Arm 2, an investigation of combination treatment of BI-1206 with rituximab, involving an initial assessment of the appropriate dose of BI-1206 that can be given in combination with rituximab (combination dose escalation cohorts).
  Interventions: Biological: Combination of BI-1206 with rituximab escalation phase
- Part B: Arm1: BI-1206 single agent expansion phase (Experimental): Part B Arm 1, an expansion cohort of up to 25 patients treated with single agent BI-1206 at the RP2D as determined in Part A Arm 1. Expansion to include a minimum of 12 chronic lymphocytic leukaemia (CLL) patients and six mantle cell lymphoma (MCL) patients.
  Interventions: Biological: BI-1206 single agent expansion phase
- Part B: Arm 2: Combination of BI-1206 with rituximab expansion phase (Experimental): Part B Arm 2, an expansion cohort of up to 25 patients treated with a combination of BI-1206 and rituximab at the RP2D as determined in Part A Arm 2. Expansion to include a minimum of 12 CLL patients and six MCL patients.
  Interventions: Biological: Combination of BI-1206 with rituximab expansion phase

INTERVENTIONS:
Biological: BI-1206 single agent dose escalation phase — BI-1206 single agent dose escalation phase to determine the MTD or maximum administered dose (MAD) and recommended Phase II dose (RP2D) for evaluation of BI-1206.
  Arms: Part A: Arm 1: BI-1206 single agent dose escalation phase
Biological: Combination of BI-1206 with rituximab escalation phase — An investigation of combination treatment of BI-1206 with rituximab.
  Arms: Part A: Arm 2: Combination of BI-1206 with rituximab escalation phase
Biological: BI-1206 single agent expansion phase — BI-1206 single agent expansion phase at the RP2D.
  Arms: Part B: Arm1: BI-1206 single agent expansion phase
Biological: Combination of BI-1206 with rituximab expansion phase — BI-1206 in combination with rituximab at the RP2D.
  Arms: Part B: Arm 2: Combination of BI-1206 with rituximab expansion phase

SUMMARY:
The purpose of this trial is to identify the tolerable dose of BI-1206 (both alone and in combination) for patients with B-cell lymphoma and leukaemia and further evaluate BI-1206 alone and in combination with an anti-CD20 antibody.

DETAILED DESCRIPTION:
The molecule CD32b is thought to be present on many B-cells including the malignant B-cells in some types of lymphoma and leukaemia. The study drug, BI-1206, is an anti-CD32b monoclonal antibody which attaches to CD32b on the surface of B-cells and is thought to act by recruiting host immune cells toward the tumour leading to cancer cell death as well as enhancing the anti-cancer effect of other anti-CD20 antibodies such as rituximab by stopping them being absorbed by cells.

The study is a first in man clinical trial of the drug called BI-1206 on its own and then also in combination with an anti-CD20 antibody (such as rituximab) which is commonly used to treat lymphoma and some types of leukaemia.

The four main aims of this trial are to find out:

* The maximum dose of BI-1206 that can be given safely to patients (to a maximum dose of 800mg) on it's own and in combination with an anti-CD20 antibody, rituximab.
* More about the potential side effects of BI-1206 and how they can be managed.
* What happens to BI-1206 inside the body.
* The effect of BI-1206 treatment (with or without rituximab) on tumour size and survival.

Approximately 81 patients with relapsed or refractory CD32b positive B-cell lymphoma or leukaemia were planned for the trial. Approximately 34 patients to establish the maximum tolerated doses (MTDs) in Part A and a further 40 to 50 patients recruited to two expansion cohorts; one of BI-1206 alone and one of BI-1206 plus rituximab (Part B). The final number depending on the number of dose escalations required to reach the MTD.

ELIGIBILITY:
Inclusion Criteria:

1. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up.
2. B-cell lymphoma or CLL proven by histology or flow cytometry, relapsed or refractory to conventional treatment, or for which no conventional therapy exists or is declined by the patient. Patients should have received at least one line of conventional previous therapy which must have included a rituximab based regimen.
3. CD32b positive malignancy as demonstrated centrally by immunohistochemistry or flow cytometry prior to study entry. Available tissue or blood must have been taken within six months of study entry.
4. Life expectancy of at least 12 weeks.
5. World Health Organisation (WHO) performance status of 0-2 (Appendix 1).
6. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week before their first dose of mAb (BI-1206 and/or rituximab) as part of this study.

   Laboratory Test Value required

   Haemoglobin (Hb) ≥9.0 g/dL (red cell support is permissible)

   Absolute neutrophil count (ANC) ≥1.0 x 10^9/L (or >0.5 x 10^9/L if due to lymphoma), granulocyte - colony stimulating factor (G-CSF) support is not permissible at screening

   Platelet count ≥50 x 10^9/L (or ≥30 x 10^9/L if due to malignant involvement of bone marrow)

   Either:

   Serum bilirubin ≤1.5 x upper limit of normal (ULN) unless raised due to Gilbert's syndrome in which case up to 3 x ULN is permissible.

   Or:

   Alanine amino-transferase (ALT) and /or aspartate amino-transferase (AST) ≤ 2.5 x ULN unless raised due to malignant hepatic involvement in which case up to 5 x ULN is permissible

   Either:

   Calculated creatinine clearance (Cockcroft Gault) ≥30 mL/min (uncorrected value)

   Or:

   Isotope clearance measurement ≥30 mL/min (corrected)
7. 18 years or over.
8. B-cell lymphoma patients only: patients has at least one measurable lesion by CT scan (defined as greater than 1.5 cm in one axis) or in the case of Waldenström's macroglobulinemia, disease must be assessable by the criteria stated in Appendix 6 of the protocol.
9. Patients recruited to Arm 2 in Parts A and B (combination arms) only: CD20 positive malignancy as demonstrated by immunohistochemistry or flow cytometry prior to trial entry.

Exclusion Criteria:

1. Allogenic bone marrow transplant within 12 months prior to the first dose of BI-1206 or presence of chronic graft versus host disease.
2. Patients with clinically active leptomeningeal or central nervous system lymphoma/leukaemia.
3. Doses of prednisolone >10 mg daily (or equipotent doses of other corticosteroids) are not permitted whilst on the study other than as pre-medication. During the screening period, doses of up to 20 mg per day may be given but the dose must be reduced to 10 mg/day by Cycle 1 Day 1 (or Day -7 in the CLL combination expansion).
4. Known or suspected hypersensitivity to study drugs.
5. Cardiac or renal amyloid light-chain (AL) amyloidosis.
6. Radiotherapy, endocrine therapy, immunotherapy, chemotherapy or investigational medicinal products during the previous 4 weeks before treatment.
7. Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 1 toxicities, which in the opinion of the Investigator and the Sponsor should not exclude the patient.
8. Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrolment and agree to use two forms of contraception (one highly effective form plus a barrier method) [oral, injected or implanted hormonal contraception and condom; intra-uterine device and condom; diaphragm with spermicidal gel and condom] or agree to sexual abstinence^4 for four weeks before entering the trial, during the trial and for twelve months after completing treatment are considered eligible.
9. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using a barrier method of contraception [condom plus spermicide] or to sexual abstinence effective from the first administration of BI-1206 or rituximab on the study, throughout the trial and for twelve months afterwards. Men with partners of child-bearing potential must also be willing to ensure that their partner uses an effective method of contraception for the same duration for example, hormonal contraception, intrauterine device, diaphragm with spermicidal gel or sexual abstinence4). Men with pregnant or lactating partners should be advised to use barrier method contraception (e.g. condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
10. Major thoracic or abdominal surgery from which the patient has not yet recovered.
11. At high medical risk because of non-malignant systemic disease including infection.
12. Known to be serologically positive for Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV).
13. Patients with an active, known or suspected autoimmune disease (not including CLL auto-immune disease). Patients with Type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger will be permitted to participate.
14. Concurrent congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA]), prior history of cardiac ischaemia or prior history of cardiac arrhythmia.
15. Patients for whom rituximab is contraindicated due to severe previous hypersensitivity or any other reason (Arm 2 in Parts A and B [combination arms] only).
16. Ongoing infection requiring treatment with antibiotics, antifungals or antivirals. Prophylactic use of antibiotics, antifungals or antivirals would not have excluded patients.
17. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.
18. Is a participant or plans to participate in another interventional clinical study, whilst taking part in this Phase I/IIa study of BI-1206. Participation in an observational study would be acceptable.
19. Current malignancies of other types, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for three years or more and are deemed at negligible risk for recurrence, are eligible for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, Prof, Principal Investigator — University of Southampton
Locations (5):
- United Kingdom (5):
  - Leicester Royal Infirmary, Leicester, England
  - Christie Hospital, Manchester, England
  - Oxford Cancer and Haematology Centre, Churchill Hospital, Oxford, England
  - Derriford Hospital, Plymouth
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial participants were enrolled at four trial sites between 27 October 2016 and 09 December 2019.
Groups:
- Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase: BI-1206 given by IV infusion to all patients once weekly for a period of four weeks, patients will then have a follow-up period of four weeks (8 week period classified as induction therapy).
  BI-1206 single agent dose escalation phase: BI-1206 single agent dose escalation phase to determine the MTD or MAD and RP2D for evaluation of BI-1206.
- Part B: Arm1: BI-1206 Single Agent Expansion Phase: Part B Arm 1, an expansion cohort of up to 25 patients treated with single agent BI-1206 at the RP2D as determined in Part A Arm 1. Expansion to include a minimum of 12 CLL patients and six MCL patients.
  BI-1206 single agent expansion phase: BI-1206 single agent expansion phase at the RP2D.
Period: Overall Study
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase
Started | 13 | 1 | 0 (Trial terminated early) | 0 (Trial terminated early)
Completed | 13 | 1 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Trial terminated before opening Part B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase | Total
Number analyzed (Participants) | 13 | 1 | 0 | 0 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  |  | 0
  Between 18 and 65 years | 5 | 1 |  |  | 6
  >=65 years | 8 | 0 |  |  | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 |  |  | 6
  Male | 8 | 0 |  |  | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 13 | 1 |  |  | 14

OUTCOME MEASURES:

1. Primary Outcome: Documenting Adverse Events (AEs), Serious Adverse Events (SAEs), Dose Limiting Toxicities (DLTs) (Graded According to NCI-CTCAE Version 4.02) and Laboratory Parameters and Determining Their Causality in Relation to BI-1206.
Description: To recommend a dose for future trials with BI-1206 by finding the highest safe dose which can be given to patients.
Time Frame: Safety data were collected from the date of written informed consent and continued for 125 days after the final administration of BI-1206 or rituximab.
Population: Safety population
Measure: Number; unit: Number of events
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase
Number analyzed (Participants) | 13 | 1 | 0 | 0
Number of events
  All AEs | 282 | 13 |  |
  Related AEs | 214 | 12 |  |
  DLT - ALT | 1 | 0 |  |
  DLT - AST | 1 | 0 |  |
  DLT - infusion related reaction | 0 | 1 |  |

2. Primary Outcome: Documenting AEs, SAEs (Graded According to NCI-CTCAE Version 4.02) and Laboratory Parameters and Determining Their Causality in Relation to BI-1206 and, Where Appropriate, Anti-CD20 Antibody.
Description: Establishing the MTD or maximum administered dose MAD of BI-1206 and an anti-CD20 antibody given once weekly for four weeks, via intravenous infusion in patients with relapsed or refractory B-cell malignancies.
Time Frame: as for outcome 1
Population: Safety population
Measure: Number; unit: BI-1206 MAD (mg)
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase
Number analyzed (Participants) | 13 | 1 | 0 | 0
BI-1206 MAD (mg) | 100 | NA — 50 mg BI-1206 given but not rituximab |  |

3. Secondary Outcome: Measurement of PK Parameter Maximum Observed Serum Concentration (Cmax) for BI-1206
Description: Maximum observed serum concentration after intravenous BI-1206 administration
Time Frame: Doses 1 and 4 (pre-infusion, end of infusion, +4, +24, +48 and +72 hours)
Population: Patients who provided serum samples before and after receiving BI-1206 for pharmacokinetic evaluation. One patient was enrolled to Part A, Arm 2 but PK parameters could not be evaluated for this patient, as there were no post-dose samples taken for the patient recruited to this cohort.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase
Number analyzed (Participants) | 12 | 0 | 0 | 0
ng/mL
  0.4 - 50 mg BI-1206 (Cohort 1, intra patient dose escalation) | 6075 [31.2 to 13100] |  |  |
  100 mg BI-1206 (Cohort 2) Dose 1 | 15600 [6990 to 19300] |  |  |
  100 mg BI-1206 (Cohort 2) Dose 4 | 12700 [8850 to 22500] |  |  |

4. Secondary Outcome: Measurement of PK Parameter Area Under the Serum Concentration-time Curve From Time 0 to the Last Time Point (AUClast) for BI-1206
Description: Area under the serum concentration-time curve from time 0 to the last time point after intravenous BI-1206 administration.
Time Frame: Doses 1 and 4 (pre-infusion, end of infusion, +4, +24, +48 and +72 hours)
Population: as for outcome 3
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase
Number analyzed (Participants) | 12 | 0 | 0 | 0
h*ng/mL
  0.4 - 50 mg BI-1206 (Cohort 1, intra patient dose escalation) | 76100 [9.1 to 384000] |  |  |
  100 mg BI-1206 (Cohort 2) Dose 1 | 462000 [129000 to 594000] |  |  |
  100 mg BI-1206 (Cohort 2) Dose 4 | 193000 [168000 to 733000] |  |  |

5. Secondary Outcome: Measurement of PK Parameter Half-life (T1/2) for BI-1206
Description: BI-1206 half-life after intravenous administration
Time Frame: Doses 1 and 4 (pre-infusion, end of infusion, +4, +24, +48 and +72 hours)
Population: as for outcome 3
Measure: Median (Full Range); unit: h
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase
Number analyzed (Participants) | 12 | 0 | 0 | 0
h
  0.4 - 2 mg BI-1206 (Cohort 1, starting dose and first intra patient escalation dose) | NA [NA to NA] — Half-life could not be assessed at these dose levels as insufficient serum concentration values were above the lower limit of detection. |  |  |
  10 - 50 mg BI-1206 (Cohort 1, intra patient dose escalation) | 17.3 [9.3 to 18.9] |  |  |
  100 mg BI-1206 (Cohort 2) Dose 1 | 16 [11.5 to 21.6] |  |  |
  100 mg BI-1206 (Cohort 2) Dose 4 | 12.1 [10.8 to 46.6] |  |  |

6. Secondary Outcome: Measurement of PK Parameter Total Body Clearance (CL) for BI-1206
Description: Total body clearance after intravenous BI-1206 administration
Time Frame: Doses 1 and 4 (pre-infusion, end of infusion, +4, +24, +48 and +72 hours)
Population: as for outcome 3
Measure: Median (Full Range); unit: mL/h/kg
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase
Number analyzed (Participants) | 12 | 0 | 0 | 0
mL/h/kg
  0.4 - 2 mg BI-1206 (Cohort 1, starting dose and first intra patient escalation dose) | NA [NA to NA] — CL could not be assessed at these dose levels as insufficient serum concentration values were above the lower limit of detection. |  |  |
  10 - 50 mg BI-1206 (Cohort 1 intra patient dose escalation) | 6.34 [2.45 to 10.8] |  |  |
  100 mg BI-1206 (Cohort 2) Dose 1 | 3.32 [1.82 to 9.63] |  |  |
  100 mg BI-1206 (Cohort 2) Dose 4 | 7.44 [6.61 to 8.64] |  |  |

7. Secondary Outcome: Measurement of PK Parameter Volume of Distribution (Vss) for BI-1206
Description: Volume of distribution after administration of BI-1206
Time Frame: Doses 1 and 4 (pre-infusion, end of infusion, +4, +24, +48 and +72 hours)
Population: as for outcome 3
Measure: Median (Full Range); unit: mL/kg
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase
Number analyzed (Participants) | 12 | 0 | 0 | 0
mL/kg
  0.4 - 2 mg BI-1206 (Cohort 1, starting dose and first intra patient escalation dose) | NA [NA to NA] — Vss could not be assessed at these dose levels as insufficient serum concentration values were above the lower limit of detection. |  |  |
  10 - 50 mg BI-1206 (Cohort 1, intra patient dose escalation) | 84.2 [60.6 to 208] |  |  |
  100 mg BI-1206 (Cohort 2) Dose 1 | 81.0 [50.5 to 182] |  |  |
  100 mg BI-1206 (Cohort 2) Dose 4 | 126 [124 to 143] |  |  |

8. Secondary Outcome: Measurement of Anti-drug Antibody (ADA) Response to BI-1206 During the BI-1206 Treatment Period Using ELISA
Description: Patients with true ADA response
Time Frame: Pre dose at weeks 1, 5 and 8, maintenance phase and off-study visit.
Population: Anti-drug antibody response population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase
Number analyzed (Participants) | 12 | 1 | 0 | 0
Participants | 0 | 0 |  |

9. Secondary Outcome: Measurement of Peripheral Blood B-lymphocyte Depletion During the BI-1206 Treatment Period Using Flow Cytometry.
Description: Number of patients with B-lymphocyte depletion during BI-1206 treatment period.
Time Frame: During induction phase (up to 8 weeks).
Population: B-lymphocyte depletion population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase
Number analyzed (Participants) | 11 | 0 | 0 | 0
Participants | 0 | 0 |  |

10. Secondary Outcome: Assessment of Best Disease Response According to Criteria for Malignant Lymphoma (Cheson, 2014) Waldenström Macroglobulinaemia Assessment Criteria (Owen 2013, Kimby 2006) or NCI Chronic Lymphocytic Leukaemia (CLL) Criteria (Hallek, 2008).
Description: To look for signs of anti-tumour activity of BI-1206 alone and in combination in patients with relapsed or refractory B-cell malignancies
Time Frame: Response evaluated 4 weeks after last dose in induction phase, every 16 weeks during maintenance phase and at off-study.
Population: Response population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase
Number analyzed (Participants) | 13 | 1 | 0 | 0
Participants
  Stable disease | 3 | 0 |  |
  Progressive disease | 7 | 0 |  |
  Not evaluable | 3 | 1 |  |

11. Secondary Outcome: Measure Progression Free Survival at 1 Year After the First BI-1206 Administration on the Study for All Patients
Description: To measure the time to disease progression and twelve month survival
Time Frame: From first BI-1206 administration up to 12 months
Population: Progression free survival population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase
Number analyzed (Participants) | 13 | 1 | 0 | 0
Participants
  Progression free & alive | 2 | 0 |  |
  Progressed, died or unknown | 11 | 1 |  |

12. Secondary Outcome: Measure Overall Survival at 1 Year After the First BI-1206 Administration on the Study for All Patients
Description: To measure the time to disease progression and twelve month survival
Time Frame: From first BI-1206 administration up to 12 months. Participants whose last reported status was not death were censored.
Population: Overall survival population
Measure: Mean (Full Range); unit: Days
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase
Number analyzed (Participants) | 5 | 0 | 0 | 0
Days | 152.2 [38 to 360] |  |  |

ADVERSE EVENTS:
Time Frame: Safety data were collected from the date of written informed consent and continued for 125 days after the final administration of BI 1206 or rituximab
Description: Trial terminated before part B opened. No patients in arm B.
Arm/Group | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase | Part B: Arm1: BI-1206 Single Agent Expansion Phase | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase
All-Cause Mortality (participants affected / at risk) | 1/13 | 0/1 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 10/13 | 1/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 13/13 | 1/1 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase (N=13) | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase (N=1) | Part B: Arm1: BI-1206 Single Agent Expansion Phase (N=0) | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase (N=0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | NA | NA
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | NA | NA
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | NA | NA
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0) | NA | NA
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | NA | NA
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | NA | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (11) | 1 (1) | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA | NA
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Arm 1: BI-1206 Single Agent Dose Escalation Phase (N=13) | Part A: Arm 2: Combination of BI-1206 With Rituximab Escalation Phase (N=1) | Part B: Arm1: BI-1206 Single Agent Expansion Phase (N=0) | Part B: Arm 2: Combination of BI-1206 With Rituximab Expansion Phase (N=0)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | NA | NA
Tachycardia (Cardiac disorders) | 4 (5) | 1 (1) | NA | NA
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | NA | NA
Cataract (Eye disorders) | 1 (1) | 0 (0) | NA | NA
Normal tension glaucoma (Eye disorders) | 1 (1) | 0 (0) | NA | NA
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | NA | NA
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | NA | NA
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Constipation (Gastrointestinal disorders) | 3 (4) | 0 (0) | NA | NA
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | NA | NA
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | NA | NA
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Lip swelling (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Nausea (Gastrointestinal disorders) | 5 (6) | 0 (0) | NA | NA
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | NA | NA
Chest discomfort (General disorders) | 1 (1) | 0 (0) | NA | NA
Chills (General disorders) | 6 (7) | 0 (0) | NA | NA
Fatigue (General disorders) | 8 (9) | 0 (0) | NA | NA
Feeling cold (General disorders) | 1 (1) | 0 (0) | NA | NA
Feeling hot (General disorders) | 2 (2) | 0 (0) | NA | NA
Non-cardiac chest pain (General disorders) | 3 (3) | 0 (0) | NA | NA
Oedema peripheral (General disorders) | 3 (3) | 0 (0) | NA | NA
Pain (General disorders) | 1 (2) | 0 (0) | NA | NA
Pyrexia (General disorders) | 5 (6) | 0 (0) | NA | NA
Folliculitis (Infections and infestations) | 2 (3) | 0 (0) | NA | NA
Lower respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0) | NA | NA
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | NA | NA
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | NA | NA
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | NA | NA
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | NA | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 9 (30) | 1 (1) | NA | NA
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | NA | NA
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | NA | NA
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | NA | NA
Blood immunoglobulin G decreased (Investigations) | 1 (1) | 0 (0) | NA | NA
Body temperature increased (Investigations) | 2 (3) | 0 (0) | NA | NA
C-reactive protein increased (Investigations) | 2 (2) | 0 (0) | NA | NA
CD4 lymphocytes decreased (Investigations) | 1 (1) | 0 (0) | NA | NA
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | NA | NA
Platelet count decreased (Investigations) | 2 (2) | 1 (1) | NA | NA
Serum ferritin increased (Investigations) | 1 (1) | 0 (0) | NA | NA
Weight decreased (Investigations) | 1 (1) | 0 (0) | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA | NA
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | NA | NA
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | NA | NA
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | NA | NA
Headache (Nervous system disorders) | 2 (6) | 0 (0) | NA | NA
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | NA | NA
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | NA | NA
Presyncope (Nervous system disorders) | 3 (4) | 0 (0) | NA | NA
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (7) | 0 (0) | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | NA
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA | NA
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA | NA
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | NA | NA
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 2 (8) | 0 (0) | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 8 (25) | 1 (2) | NA | NA
Flushing (Vascular disorders) | 5 (12) | 0 (0) | NA | NA
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | NA | NA
Hypertension (Vascular disorders) | 4 (8) | 0 (0) | NA | NA
Hypotension (Vascular disorders) | 6 (11) | 1 (1) | NA | NA
Pallor (Vascular disorders) | 1 (1) | 0 (0) | NA | NA
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | NA | NA

LIMITATIONS AND CAVEATS:
The trial was terminated early by the Sponsor based on a strategic decision and not a safety related decision. At the time of trial termination, 14 patients had received BI-1206. No patients received rituximab. As a result of the early termination Part B of the trial did not open.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT02933320/Prot_SAP_000.pdf